CLINICAL TRIAL: NCT05872919
Title: Telehealth and Challenges in Statin Adherence in Patients With Diabetes: A Randomized Controlled Trial
Brief Title: Telenhealth and Adherence to Stains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amna A. Desouky, MD, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Adherence for medication
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Telehealth , Lipid Lowering Medication Adherence

STUDY DESIGN:
Intervention Model Description: Eligible patients will be offered to participate. Willing patients will be randomly assigned to one of two groups: Two arms study design: first arm (control group)won't receive intervention while the second arm (intervention group) will receive telenursing intervention through SMS; Is a text messages will be sent to the intervention group comprised of a reminder on when, how to take lipid lowering medication, benefits, and adverse effect of not taken the drug as prescribed for three months duration. SMS (Short Messaging Service) will be sent three times per week in the first six weeks and twice per week in the second six weeks.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: MA will provide randomization AD will assess participant at baseline and follow-up EH will deliver the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): will not receive the intervention
- Study group (Experimental): will receive the intervention
  Interventions: Other: SMS reminder massages about adherence

INTERVENTIONS:
Other: SMS reminder massages about adherence — SMS three-times per week in the first six weeks and twice per week in the second six weeks reminding the patient about adherence to prescribed medication
  Arms: Study group

SUMMARY:
To evaluate the effect of telehealth through short messaging services (SMSs) on adherence to statins in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Both sexes
* Type 1 and 2 diabetes
* Had a prescription of lipid lowering medication with a minimum duration of two weeks
* Have an active contact phone number that can receive text messages
* Able to read SMS text messages (patient, or family member)

Exclusion criteria:

* Communication impairment
* Taking any psychotropic medications
* Familial hypercholesterolemia
* Already established coronary heart disease
* not on lipid lowering medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Adherence rate | 6 and 12 weeks
  Adherence rate was measured by:
  1. Pill counting (PC) Pill count (PC) Is an objective mesearrment, calculated by the sum of days covered by lipid-lowering medication divided by the number of days in that period.
  Investigators calculated the index date for adherence on the day of recruitment for each patient.
  Patients were considered to have good adherence to lipid-lowering medication if their estimated PC was ≥80%,
  Equation : Sum of days covered by lipid-lowering medication / number of days in that period × 100.
  Percentage ≧ 80% means a good medication adherence
  Percentage < 80% means a poor medication adherence
Adherence rate | 6 and 12 weeks
  Medication Adherence Reporting Scale -5 (MARS-5) is a self-reporting scale. Is a subjective method of mesearrment, It is a 5 five-point Likert scale response ranging from 1 (always) to 5 (never).
  The total score of the MARS-5 ranges from 5 to 25
  Mean score ≥20 means good medication adherence
  Mean score < 20 means poor medication adherence

SECONDARY OUTCOMES:
Lipid profile | at 12 week
  Mean score of lipid profile will be monitored at follow up times comparison between baseline and follow up measurements will be done
Acute cardiovascular events (CVE) | at 12 weeks
  Number of cases who will be hospitalized or exposed to acute cardiovascular events (CVD) within follow periods.
Mortality | at 12 weeks
  Number of death or mortality within follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt